CLINICAL TRIAL: NCT07097584
Title: Effect of Small Double-lumen Tube on the Intubation Time of Thoracoscopic Pulmonectomy in Asian Women: a Randomized Controlled Clinical Trial
Brief Title: Effect of Small Double-lumen Tube on the Intubation Time of Thoracoscopic Pulmonectomy in Asian Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Gu Bin, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-2025-841
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Women; Asian; Thoracic Surgery With One-lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologists do not implement the blinding method for the patient grouping, while the physicians conducting the postoperative follow-up implement the blinding method for the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Down-size Left Double-lumen Endobronchial Tube Group (Experimental)
  Interventions: Device: Selecting the size of a Left Double-lumen endobronchialtube one size smaller than the traditional method
- The Regular Left Double-lumen Endobronchial Tube Group (Active Comparator)
  Interventions: Device: Selecting the size of a Left Double-lumen endobronchialtube according to traditional methods

INTERVENTIONS:
Device: Selecting the size of a Left Double-lumen endobronchialtube one size smaller than the traditional method — During tracheal intubation，choose a Left Double-lumen Endobronchial Tubethat is one size smaller than the traditional method.In this study, all patients planned to be enrolled are female. In experimental group the relationship between height and size is roughly as follows: For patients with a height between 152 - 165 cm, a 32Fr (French) tube is often selected. For patients with a height between 165 - 177 cm, a 35Fr tube is often selected. For patients with a height of more than 177 cm, a 37Fr tube is often selected.
  Arms: The Down-size Left Double-lumen Endobronchial Tube Group
Device: Selecting the size of a Left Double-lumen endobronchialtube according to traditional methods — During tracheal intubation，choose the regular Left Double-lumen endobronchial tube according to the traditional method. The selection of double-lumen tube sizes using traditional methods relies on two factors: height and gender. In this study, all patients planned to be enrolled are female, so the traditional corresponding relationship is roughly as follows:
  For patients with a height of less than 152 cm, a 32Fr (French) tube is often selected.
  For patients with a height between 152 - 165 cm, a 35Fr tube is often selected. For patients with a height between 165 - 177 cm, a 37Fr tube is often selected. For patients with a height of more than 177 cm, a 39Fr tube is often selected.
  Arms: The Regular Left Double-lumen Endobronchial Tube Group

SUMMARY:
The purpose of this experiment is to verify whether selecting a double-lumen tube one size smaller based on the traditional personalized method can shorten the intubation time without increasing ventilation complications when performing tracheal intubation for thoracic surgery in Asian women.Patients receive double-lumen tubes of a size selected based on the traditional personalized method or one size smaller than that chosen by the traditional method during tracheal intubation. The primary outcome is the time duration required to complete Double-lumen tube intubation and positioning.

DETAILED DESCRIPTION:
The selection of double-lumen tube sizes using traditional methods relies on two factors: height and gender. In this study, all patients planned to be enrolled are female, so the traditional corresponding relationship is roughly as follows: For patients with a height of less than 152 cm, a 32Fr (French) tube is often selected. For patients with a height between 152 - 165 cm, a 35Fr tube is often selected. For patients with a height between 165 - 177 cm, a 37Fr tube is often selected. For patients with a height of more than 177 cm, a 39Fr tube is often selected.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoscopic pulmonary resection using a left double-lumen tube under general anesthesia.
* Patients aged 18-80 years
* Chest CT scan in our hospital within one month before surgery
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Anticipated difficult airway
* Patients with tracheal/left main bronchus anomalies
* Height <152 cm
* Refused to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intubation allocation time | During induction of general anesthesia
  The time duration required to complete Double-lumen tube intubation and positioning

SECONDARY OUTCOMES:
Time of laryngoscope insertion | During induction of general anesthesia
Time of double-lumen tube insertion | During induction of general anesthesia
  Under videolaryngoscopy，the LDLT (left double-lumen tube) with the stylet is introduced into the glottis with the tip oriented anteriorly. After the bronchial cuff passes through the glottis the stylet is removed and the tube is rotated 90 degrees counterclockwise.The LDLT is then advanced to the predicted depth: LDLT depth (cm) = 12 + [patient height (cm) × 10-¹]Intubation time is defined as the period from insertion of the laryngoscope blade to completion of LDLT placement.
Time of successfully positioning of fiberoptic bronchoscope in supine position | During induction of general anesthesia
  Following intubation, the attending anesthesiologist inserted the fiberoptic bronchoscope (FOB) to reposition the left-sided double-lumen tube (LDLT) for optimal placement.（Confirmed by FOB: The left upper lobe and lower lobe bronchi were clearly visualized through the bronchial lumen, the left mainstem bronchus was seen via the tracheal lumen, and the bronchial cuff was positioned just below the carina).
First-pass success rate of intubation | During induction of general anesthesia
  Fiberoptic bronchoscopic adjustment immediately following intubation，if the DLT moves less than 1.0cm after the first intubation, it is regarded as successful
Number of intubation attempts | During induction of general anesthesia
The incidence of Intubation difficulty | During induction of general anesthesia
  Intubation difficulty（when an anesthetist with over 3 years of DLT intubation experience needs ≥3 attempts or intubation time ≥10 min during DLT intubation）
The incidence of air leakage in double-lumen bronchial tubes | During induction of general anesthesia
  After inflating the endotracheal tube cuff with 2-6 ml of air and the bronchial cuff with 1-3 ml of air respectively, cuff pressures are measured and should be < 25 cm H₂O and < 20 cm H₂O respectively. Absence of an air leak from the endotracheal tube when peak airway pressure reaches 30 cm H₂O during positive-pressure ventilation is considered an indicator of adequate seal.
Videolaryngoscope VIDIAC score | During induction of general anesthesia
  The VIDIAC score is comprised of: E, the interaction between the blade tip and epiglottis; V, the best view of the vocal cords from the blade camera; and A, enlargement of the arytenoids. The score range of the VIDIAC score is from -1 to 5 points. The VIDIAC score classification is as follows: Easy, with a score of -1 or 0; Moderate, with a score of 1; Difficult, with a score of 2; Severe, with a score of ≥3.
Intubation resistance | During induction of general anesthesia
  Intubation Resistance
  1. No resistance
  2. Mild resistance
  3. Moderate resistance (Significant resistance encountered at the subglottis, although the tracheal tube segment can be advanced past the subglottis)
  4. Severe resistance(The tracheal tube segment cannot pass the subglottis and must be replaced with the next smaller size)
Intubation depth | During induction of general anesthesia
  LDLT depth (cm) = 12 + [patient height (cm) × 10-¹
Adverse events during intubation | During induction of general anesthesia
Misplacement rate after position change (movement distance>1.0 cm) | During induction of general anesthesia
  if the DLT moves more than 1.0cm after the first intubation, it is regarded as Misplacement
Campos atelectasis classification | 5 minutes and 20 minutes after the distal port of the double-lumen tube is opened
  Campos Classification of Lung Collapse:
  Excellent: The operated lung is completely collapsed, the surgical field is satisfactorily exposed, and no intervention by the surgeon is required.
  Good: The operated lung is mostly collapsed with some residual gas in the lung, but there is no ventilation in the lung, and the surgical field is relatively satisfactorily exposed.
  Poor: The operated lung is not collapsed or only partially collapsed, which interferes with the surgical operation and requires intervention by the surgeon.
Accumulated usage times of fiberoptic bronchoscope | During the operation
  SaO₂≤90% and ≥1min, airway pressure>35cm H₂O, poor lung atelectasis, or according to experience, all need to use fiberoptic bronchoscope to confirm the position
The incidence of misplacement during the operation | during the operation
  if the DLT moves more than 1.0cm after the first intubation, it is regarded as Misplacement
Number of intraoperative double-lumen tube adjustments | During the operation
The incidence of hypoxemia intraoperatively | During the operation
  hypoxemia means arterial oxygen saturation≤90%, and ≥60s
Intraoperative single-lung ventilation time | through study completion，an average of 1-4 hours
Carina mucosa injury score | During the operation
  after repositioning to supine position, the double-lumen tube is withdrawn to the main trachea, and the mucosa within a 1cm radius of the carina is assessed using a fiberoptic bronchoscope
Multiplanar Reconstruction（MPR) of lung CT measurement data | after operation，an average of 1-3 days
  Left main bronchus transverse diameter (TD-LMB) (cm) Left main bronchus anteroposterior diameter (APD-LMB) (mm) Left main bronchus equivalent diameter (ED-LMB) (cm) DLT model selected based on MPR
Bronchial window measurement data | after operation，an average of 1-3 days
  Bronchial window measurement data Left main bronchus anteroposterior diameter (APD-LMB) (mm) DLT model selected based on bronchial window
PACU stay time | after operation，an average of 60-120 minutes
The incidence of sore throat | One hour, twenty-four hours, forty-eight hours after surgery
The incidence of postoperative cough | One hour, twenty-four hours, forty-eight hours ，thirty days after surgery
Postoperative pain score | twenty-four hours, forty-eight hours ，thirty days after surgery
  The Numeric Rating Scale (NRS) is a widely used tool for assessing pain intensity, recognized for its simplicity, ease of administration, and high reliability across various patient populations.
  The scale ranges from 0 to 10, where:
  0 indicates "no pain at all." 10 represents "the worst imaginable pain."
Postoperative chest tube removal time | after operation through study completion，an average of 3-4 days
Length of hospital stay after surgery | after operation through study completion，an average of 3-7 days
Postoperative 30-day complications | within 30 days after surgery
  Postoperative 30-day complications by using Clavien-Dindo score
The incidence of postoperative pulmonary complications | within 30 days after surgery
  postoperative pulmonary complications include: Pneumonia,Atelectasis,Respiratory failure,Pleural effusion,Bronchospasm,Pulmonary embolism If any of the above conditions is present, it is considered that there is a postoperative pulmonary complication.
the postoperative recovery | on postoperative day 1
  The postoperative recovery is assessed using the quality of recovery-15 questionnaire (QoR-15) .The QoR-15 has 15 questions. Each question is rated on a 10-point scale, ranging from 0 (none of the time or poor) to 10 (all of the time or excellent). The maximum score (best recovery) is 150
heart rate before and after intubation | Baseline. At 1，2,5 minutes after intubation.
mean arterial pressure before and after intubation | baseline.At 1，2,5 minutes after intubation.
Intraoperative Partial Pressure of Arterial Oxygen (PaO₂) | During the operation
  arterial blood can be drawn from the specimen for examination.
Intraoperative Partial Pressure of Arterial Carbon Dioxide (PaCO₂) | During the operation
  arterial blood can be drawn from the specimen for examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
We will share data on ClinicalTrials.gov, and data sharing will be always available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: starting about 6 months after publication